CLINICAL TRIAL: NCT04550819
Title: Prevention of Duodenobiliary Reflux Via Intraintestinal Extended Biliary Stents in Patients With Biliary Stricture
Brief Title: Intraintestinal Extended Biliary Stents Preventing Duodenobiliary Reflux in Patients With Biliary Stricture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Huang Yonghui, Chief physician, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: X20200703
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Bile Duct Stricture

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IEBSs in malignant extrahepatic biliary stricture (Experimental): Intraintestinal extended biliary stents(IEBSs) in patients with malignant extrahepatic biliary stricture
  Interventions: Procedure: intraintestinal extended biliary stents
- CPBSs in malignant extrahepatic biliary stricture (Active Comparator): Conventional plastic biliary stents(CPBSs) in patients with malignant extrahepatic biliary stricture
  Interventions: Procedure: ordinary plastic biliary stents
- IEBSs in benign extrahepatic biliary stricture (Experimental): Intraintestinal extended biliary stents(IEBSs) in patients with benign extrahepatic biliary stricture
  Interventions: Procedure: intraintestinal extended biliary stents
- CPBSs in benign extrahepatic biliary stricture (Active Comparator): Conventional plastic biliary stents(CPBSs) in patients with benign extrahepatic biliary stricture
  Interventions: Procedure: ordinary plastic biliary stents

INTERVENTIONS:
Procedure: intraintestinal extended biliary stents — The test group will be placed intraintestinal extended biliary stents in intrahepatic bile duct in ERCP
  Arms: IEBSs in benign extrahepatic biliary stricture; IEBSs in malignant extrahepatic biliary stricture
Procedure: ordinary plastic biliary stents — The test group will be placed ordinary plastic biliary stents in intrahepatic bile duct in ERCP
  Arms: CPBSs in benign extrahepatic biliary stricture; CPBSs in malignant extrahepatic biliary stricture

SUMMARY:
Metal or plastic biliary stents placement under Endoscopic Retrograde Cholangiopancreatography(ERCP) is a well-established treatment for patients with benign biliary obstruction to relieve jaundice, a palliative treatment for patients with unresectable malignant pancreaticobiliary obstruction and a bridge to surgery for patients with resectable disease. The main limitation of long time plastic stents is stents occlusion. Biliary plastic stents are changed every 2 to 3 months due to an expected median patency from 77 to 126 days.Metal stents present a lower risk of recurring biliary occlusion, yet high cost and stents occlusion are eventually inevitable. The mechanism of biliary stents occlusion include biliary sludge of the accumulation of bacteria and duodenal biliary reflux .The anti-reflux barrier of Oddi's sphincter disappears after the insertion of biliary stents and the pressure in bile duct lowers the duodenale, which cause the retrograde flow of duodenal material into the biliary ducts. Besides, ordinary biliary plastic stent is short which can also shortens the length of duodenal biliary reflux . Therefore, trying to prevent the duodenal biliary reflux is very important in reducing biliary stents occlusion and it is gradually concerned by clinical researchers. Some studies have showed that plastic stents with antireflux valves can effectively reduce the biliary stent stricture and prolong the stents patency, which means reducing duodenobiliary reflux is surely useful for keeping biliary stent patency.So,we assume to explore an innovatively intraintestinal extended biliary stents (reformed with nasobiliary tube ) as substitution for ordinary biliary plastic stent to prevent the duodenobiliary reflux by extending the length of duodenal content reflux and avoid the stents shift via suspending in intrahepatic duct. In this study,we will design a multicenter stratified randomized controlled trial to compare the patency of intraintestinal extended biliary stents and ordinary plastic biliary stents in patients with malignant or benign biliary obstruction respectively and evaluate the effect of intraintestinal extended biliary stents for the prevention of duodenobiliary reflux.

DETAILED DESCRIPTION:
Metal or plastic biliary stents placement under ERCP is a well-established treatment for patients with benign biliary obstruction to relieve jaundice, a palliative treatment for patients with unresectable malignant pancreaticobiliary obstruction and a bridge to surgery for patients with resectable disease. Single or multiple plastic stents are recommended for patients with benign stricture of the common bile duct or malignant stricture if the expected survival is less than 4 months. The main limitation of long time plastic stents is stents occlusion. Biliary plastic stents are changed every 2 to 3 months due to an expected median patency from 77 to 126 days.Metal stents present a lower risk of recurring biliary occlusion, yet high cost and stents occlusion are eventually inevitable. The mechanism of biliary stents occlusion include biliary sludge of the accumulation of bacteria and duodenal biliary reflux .The anti-reflux barrier of Oddi's sphincter disappears after the insertion of biliary stents and the pressure in bile duct lowers the duodenale, which cause the retrograde flow of duodenal material into the biliary ducts. Besides, ordinary biliary plastic stent is short which can also shortens the length of duodenal biliary reflux . Therefore, trying to prevent the duodenal biliary reflux is very important in reducing biliary stents occlusion and it is gradually concerned by clinical researchers. Some studies have showed that plastic stents with antireflux valves can effectively reduce the biliary stent stricture and prolong the stents patency, which means reducing duodenobiliary reflux is surely useful for keeping biliary stent patency.So,we assume to explore an innovatively intraintestinal extended biliary stents with length of 26cm (reformed with nasobiliary tube ) as substitution for ordinary biliary plastic stent to prevent the duodenobiliary reflux by extending the length of duodenal content reflux and avoid the stents shift via suspending in intrahepatic duct. In this study,we will design a multicenter stratified randomized controlled trial to compare the patency of intraintestinal extended biliary stents and ordinary plastic biliary stents in patients with malignant or benign biliary obstruction respectively and evaluate the effect of intraintestinal extended biliary stents for the prevention of duodenobiliary reflux.

This prospective study will be performed at 6 tertiary hospitals in China.The investigators will recruit patients according to admission criteria and exclusion criteria.The patients stratified by malignant and benign biliary obstruction will be randomized (at a 1:1 ratio) to intraintestinal extended biliary stents group (experimental group) and ordinary plastic biliary stents group (control group).The experimental groups will be placed the intraintestinal extended biliary stents in intrahepatic bile duct in ERCP. The control group will be placed ordinary plastic biliary stents in ERCP. The primary endpoint is the duration of stent patency and the rate of stent occlusion.The secondary outcomes include the mortality of each group、adverse events and the rate of technical success.

ELIGIBILITY:
Inclusion Criteria:

* Malignant or benign extrahepatic biliary stricture,available for insertion of biliary stents in ERCP to alleviate biliary stricture

Exclusion Criteria:

* Patients with malignant or benign biliary stricture do not agree with endoscopic treatment
* Patients agree with metal biliary stents
* Patients with resectable biliary occlusion
* A guidewire could not be passed through the stricture
* Patients with an expected life survival <3months
* Patients with duodenal obstruction and duodenal endoscopy could not be reached to papillary

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 724 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
the duration of stent patency and stent occlusion rate | 12 months after ERCP
  Patients with symptoms of cholangitis and worsening liver function tests suggestive of cholestasis are considered as premature stent occlusion.

SECONDARY OUTCOMES:
mortality of each group | 12 months after ERCP
  We will compare the mortality of each group after the insertion of biliary stents.
adverse events | 12 months after ERCP
  Adverse events include complications of post ERCP such as pancreatitis,biliary infection, bleeding, perforation，and stent migration
the rate of technical success | 12 months after ERCP
  Technical success is defined as successful insertion of the stent into the bile duct during ERCP

CONTACTS AND LOCATIONS:
Overall Officials: Yonghui Huang, archiater, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dumonceau JM, Tringali A, Blero D, Deviere J, Laugiers R, Heresbach D, Costamagna G; European Society of Gastrointestinal Endoscopy. Biliary stenting: indications, choice of stents and results: European Society of Gastrointestinal Endoscopy (ESGE) clinical guideline. Endoscopy. 2012 Mar;44(3):277-98. doi: 10.1055/s-0031-1291633. Epub 2012 Feb 1. PMID 22297801
- [Background] Libby ED, Leung JW. Prevention of biliary stent clogging: a clinical review. Am J Gastroenterol. 1996 Jul;91(7):1301-8. PMID 8677983
- [Background] van Berkel AM, Boland C, Redekop WK, Bergman JJ, Groen AK, Tytgat GN, Huibregtse K. A prospective randomized trial of Teflon versus polyethylene stents for distal malignant biliary obstruction. Endoscopy. 1998 Oct;30(8):681-6. doi: 10.1055/s-2007-1001388. PMID 9865556
- [Background] van Berkel AM, Bruno MJ, Bergman JJ, van Deventer SJ, Tytgat GN, Huibregtse K. A prospective randomized study of hydrophilic polymer-coated polyurethane versus polyethylene stents in distal malignant biliary obstruction. Endoscopy. 2003 Jun;35(6):478-82. doi: 10.1055/s-2003-39666. PMID 12783344
- [Background] Reddy DN, Banerjee R, Choung OW. Antireflux biliary stents: are they the solution to stent occlusions? Curr Gastroenterol Rep. 2006 Apr;8(2):156-60. doi: 10.1007/s11894-006-0012-x. PMID 16533479
- [Background] van Berkel AM, van Marle J, van Veen H, Groen AK, Huibregtse K. A scanning electron microscopic study of biliary stent materials. Gastrointest Endosc. 2000 Jan;51(1):19-22. doi: 10.1016/s0016-5107(00)70380-4. PMID 10625789
- [Background] Groen AK, Out T, Huibregtse K, Delzenne B, Hoek FJ, Tytgat GN. Characterization of the content of occluded biliary endoprostheses. Endoscopy. 1987 Mar;19(2):57-9. doi: 10.1055/s-2007-1018235. PMID 3106022
- [Background] Speer AG, Cotton PB, Rode J, Seddon AM, Neal CR, Holton J, Costerton JW. Biliary stent blockage with bacterial biofilm. A light and electron microscopy study. Ann Intern Med. 1988 Apr;108(4):546-53. doi: 10.7326/0003-4819-108-4-546. PMID 2450501
- [Background] Liu YF, Saccone GT, Thune A, Baker RA, Harvey JR, Toouli J. Sphincter of Oddi regulates flow by acting as a variable resistor to flow. Am J Physiol. 1992 Nov;263(5 Pt 1):G683-9. doi: 10.1152/ajpgi.1992.263.5.G683. PMID 1443142
- [Background] Donelli G, Guaglianone E, Di Rosa R, Fiocca F, Basoli A. Plastic biliary stent occlusion: factors involved and possible preventive approaches. Clin Med Res. 2007 Mar;5(1):53-60. doi: 10.3121/cmr.2007.683. PMID 17456835
- [Background] van Berkel AM, van Marle J, Groen AK, Bruno MJ. Mechanisms of biliary stent clogging: confocal laser scanning and scanning electron microscopy. Endoscopy. 2005 Aug;37(8):729-34. doi: 10.1055/s-2005-870131. PMID 16032491
- [Background] Dua KS, Reddy ND, Rao VG, Banerjee R, Medda B, Lang I. Impact of reducing duodenobiliary reflux on biliary stent patency: an in vitro evaluation and a prospective randomized clinical trial that used a biliary stent with an antireflux valve. Gastrointest Endosc. 2007 May;65(6):819-28. doi: 10.1016/j.gie.2006.09.011. Epub 2007 Mar 26. PMID 17383650
- [Background] Vihervaara H, Gronroos JM, Hurme S, Gullichsen R, Salminen P. Antireflux Versus Conventional Plastic Stent in Malignant Biliary Obstruction: A Prospective Randomized Study. J Laparoendosc Adv Surg Tech A. 2017 Jan;27(1):53-57. doi: 10.1089/lap.2016.0178. Epub 2016 Oct 18. PMID 27754790
- [Background] Yang F, Ren Z, Chai Q, Cui G, Jiang L, Chen H, Feng Z, Chen X, Ji J, Zhou L, Wang W, Zheng S. A novel biliary stent coated with silver nanoparticles prolongs the unobstructed period and survival via anti-bacterial activity. Sci Rep. 2016 Feb 17;6:21714. doi: 10.1038/srep21714. PMID 26883081